**Study Title**: Delivering Health: An Integrated Approach to Address Diabetes in

the Context of Food Insecurity

**Principal Investigator**: Krista Langston

University of Arkansas for Medical Sciences Northwest 2708 S. 48<sup>th</sup> Street

2708 S. 48<sup>th</sup> Street Springdale, AR 72762 Telephone: 479-713-8691 Email: KLangston@uams.edu

**Study location**: University of Arkansas for Medical Sciences Northwest

4301 West Markham Street Little Rock, AR 72205

Version #: 10
Date: 20230222

IRB#260304
Page 1

Insecurity

PI: Krista Langston

## **Background and Rationale**

Decades of increasing incidence of type 2 diabetes (T2D) present a multifaceted challenge to the health of a growing number of Americans, affecting their diets and how they live life. Approximately 30 million (~9%) of all people in the US have T2D. 1 and this number is expected to continue to rise. It is estimated that the prevalence will increase to more than 54 million Americans by 2030.<sup>2</sup> At the same time, 15 million (11.8%) US households experience food insecurity, which is associated with risk for T2D and other chronic diseases. Both T2D and food insecurity are even more prevalent in Arkansas, with rates of T2D and food insecurity at 12.2%<sup>5</sup> and 17.3%, <sup>6</sup> respectively. T2D and food insecurity are strongly associated for U.S. adults: Very low food security is associated with an over 100% increase in prevalence of T2D compared with adults from high food-secure households. Even for adults in marginally food secure households, probability of T2D increases by 59%.4

~40 million Americans are food insecure,<sup>3</sup> and food insecurity is associated with double the prevalence of T2D.<sup>4</sup> Food insecure people face many risk factors for unmanaged T2D,<sup>7</sup> including poor diet quality.<sup>8-12</sup> insufficient physical activity.<sup>13-15</sup> and lack of access to health care.<sup>16-18</sup> Unmanaged T2D can lead to increased risk of serious complications, including neuropathy, nephropathy, retinopathy, atherosclerosis, heart attack, stroke, and death. 19

~46 million Americans per year turn to food pantries and related programs to help meet household nutritional needs.<sup>20</sup> An estimated 33% of food pantry client households have at least one member with T2D.<sup>20</sup> Among these, 46% use food pantries at least six times per year.<sup>21</sup>

However, food pantries are not a long-term solution to improve health for food insecure people with T2D. Most food pantries do not provide food of sufficient dietary quality to support a healthy lifestyle, particularly for vitamins A and C and calcium. <sup>22</sup> Current food pantry clients' diet quality is insufficient for caloric intake, fruits, vegetables, and dairy.<sup>23</sup>

Diabetes self-management education (DSME) is an approach with documented efficacy in helping people manage T2D. DSME supports informed decision-making, encourages goal setting and problem solving, and improves self-care behaviors.<sup>24</sup> Across many populations, DSME improves glycemic control;<sup>25</sup> lowers body mass index (BMI);<sup>26</sup> improves diabetes knowledge,<sup>27</sup> diet quality, <sup>28</sup> physical activity, <sup>29</sup> and self-efficacy; <sup>27</sup> reduces health care costs and hospitalizations. 30,31 and increases use of primary care and preventive services. 32

Recent studies have shown promise for DSME among food pantry clients with T2D. One study paired DSME classes with T2D-appropriate food boxes distributed at food banks and found significant improvements in glycemic control.<sup>33</sup> However, this study suffered from problems with attendance and retention, retaining only 42% of participants. In a follow-up trial, only 20% engaged fully with the DSME and food box intervention (i.e., picked up  $\geq 9$  of 11 food distributions, attended 2 DSME classes, etc.).<sup>34</sup>

By removing barriers to attendance and retention, our research team will leverage the full potential of home-delivered T2D-appropriate food boxes paired with DSME. We have

IRB#260304 Version #: 10 Date: 20230222

PI: Krista Langston

successfully adapted diabetes education for delivery in community settings, including homes, faith-based organizations, and community centers.<sup>35</sup> We have adapted DSME for people from diverse cultural backgrounds who face economic, transportation, health care, and health literacy barriers.<sup>36</sup> We are experienced at developing interventions to improve health of low-income food insecure people, including food pantry interventions to improve access to healthy food.<sup>37,38</sup>

We propose a study to develop and evaluate the efficacy of a plain-language DSME curriculum to improve the nutritional health, physical activity, and health outcomes of low-income food insecure people with T2D. We will home-deliver this curriculum along with T2D-appropriate healthy food boxes to mitigate difficulties associated with access to healthy food and attendance at DSME sessions outside of the home. We hypothesize that this approach will lead to improvements in participants' glycemic control, diet quality, and other outcomes.

## **Objective**

Develop, implement, and evaluate the effectiveness of an intervention to use home-delivery of T2D-appropriate food boxes with plain language adapted education materials, in English, Spanish, and Marshallese, to improve the nutritional health, physical activity, and health outcomes of low-income food insecure people with T2D.

## **Study Design and Procedures**

**Stakeholder involvement** Stakeholders were involved in problem selection and project development. Stakeholders will participate in adapting the DSME curriculum. To ensure the study captures outcomes important to each stakeholder group, stakeholders helped choose study outcomes. Stakeholders will be invited to help interpret study results and to participate in dissemination as co-authors of manuscripts, reports, and presentations.

Project activities 1. Adapt DSME curriculum for use by low-income food insecure

communities. As part of the development, we will incorporate T2D-appropriate recipes and information on cooking and shopping when on a limited budget and with foods commonly found at food pantries. In addition, 12 videos will be created and posted on a freely accessible UAMS website to introduce and reinforce key DSME concepts.

## **Table 1. 12-week Adapted ACP Curriculum Modules**

- 1. What is Diabetes?
- 2. Healthy Eating Part 1Healthy
- 3. Healthy Eating Part 2
- 4. Physical Activity Part 1
- 5. Physical Activity Part 2
- 6. Monitoring Diabetes
- 7. Acute Complications
- 8. Chronic Complications Part 1
- 9. Chronic Complications Part 2
- 10. Medication Management
- 11. Healthy Coping
- 12. Problem Solving

PI: Krista Langston

The 12 adapted modules are presented in **Table 1**. In the study, these modules will be delivered to the participants on paper in the T2D-appropriate food boxes and in easy to access online versions, which link to the videos summarizing the key concepts and demonstrating cooking techniques. All materials are translated into English, Spanish, and Marshallese.

<u>2. Design T2D-appropriate food boxes.</u> The project team led by an endocrinologist, registered nurse, and registered dietitian designed 12 weekly food boxes to be home delivered to each participant. The boxes were adapted from the American Diabetes Association Create Your Plate method,<sup>49</sup> which emphasizes non-starchy vegetables, proteins, and grains, consistent with the meal pattern promoted in the ACP DSME.<sup>48</sup> In addition, the boxes will include food that largely reflects Feeding America's Foods to Encourage framework,<sup>50</sup> which was developed by nutrition experts and food bank leaders to meet USDA dietary guidelines<sup>51</sup> and MyPlate framework.<sup>52</sup>

The boxes will include ~9,000 calories of food, equivalent to the amount the average household would receive <u>pro-rated per week</u> from an average Arkansas food pantry.<sup>37</sup> Each box will include fresh fruits and vegetables, as well as the ingredients necessary to prepare the recipes included with that week's DSME curriculum. If a certain item is unavailable or out of stock, there is a list of potential substitutions that are of equal nutritional content compared to the first

choice food item. Each week's box will include an educational fact sheet of the week's DSME module. including links and OR codes leading to the videos. Links to the week's online materials, which present the same content as the paper materials, will be texted or emailed to each participant based on their preferred contact method on the day each box is delivered. Table 2 shows an example T2Dappropriate food box.

3. Recruit and enroll up to 110 participants. Study participants may be

| Table 2. Example of T2DM-appropriate Food Box | |
|---|---|
| Fruit | <ul> <li>1- 20 oz. Canned Pineapple Tidbits in Natural<br/>Juice</li> </ul> |
| | 1- 15 oz. Canned Lite Sliced Peaches |
| | 3 Fresh Apples |
| Vegetables | <ul> <li>1- 15 oz. Canned Mixed Vegetables</li> </ul> |
| | <ul> <li>1- 14.5 oz. Canned No Salt Added Green</li> </ul> |
| | Beans |
| | <ul> <li>2 Fresh Sweet Potatoes</li> </ul> |
| | <ul> <li>1 Fresh Onion</li> </ul> |
| | <ul> <li>1- 10 oz. bag Frozen Spinach</li> </ul> |
| Meat/Protein | <ul> <li>1- 15 oz. can No Salt Added Black Beans</li> </ul> |
| | <ul> <li>1- 10 oz. Canned Chicken</li> </ul> |
| | <ul> <li>1- 12 oz. Canned Tuna</li> </ul> |
| | <ul> <li>1- Dozen Large Eggs</li> </ul> |
| Whole | 1- 10 count Whole Wheat Tortillas |
| Grains | <ul> <li>1- 14 oz. box Instant Brown Rice</li> </ul> |
| Dairy | 1- Gallon 1% Milk |
| | <ul> <li>1- 10 oz. bag Part Skim Mozzarella String</li> </ul> |
| | Cheese |
| Other | <ul> <li>1-8 fl oz. bottle Extra Virgin Olive Oil (this is</li> </ul> |
| | included in the calorie count) |

recruited from waiting areas of food pantries located in Benton and Washington Counties in northwest Arkansas. (See Letters of Support from local food pantries.) Due to social distancing and public health guidelines related to COVID-19 each of the food pantries have established drive-thru clinics where participants can remain isolated in their vehicles while completing data collection. Participants may use these drive-thru clinics for consent and all biometric collection.

PI: Krista Langston

If COVID-19 regulations are lifted and food pantries are welcoming clients inside, consent and biometrics will be collected in a private area of the facility. In our preliminary data from 247 food pantry clients, 95% of clients in this region screen positive for food insecurity, and ~30% report at least one household member diagnosed with T2D. Participant inclusion criteria include: report food insecurity (confirmed by adapted 10-item screener<sup>53</sup>); 18 years of age or older; report T2D (confirmed by having an HbA1c equal to or greater than 7 at initial data collection immediately following consent. Participant exclusion criteria include conditions making it unlikely the participant will be able to follow the protocol, such as terminal illness, non-ambulatory, severe mental illness, severely impaired vision or hearing, eating disorder, pregnant, or plans to move out of the geographic region. Only one adult per household will be enrolled. Individuals under 18 years old are not included in the proposed study because the intervention is designed for adults with T2D.

Consent materials will be available in English, Spanish, or Marshallese and will use plain language. Eligible participants will be provided a copy of the consent to review, and participants will have the opportunity to ask questions, consent, and enroll in the study. The consent process will include providing information to the potential participants and the opportunity to have bilingual Marshallese or Spanish speaking staff answer questions regarding study participation. The consent document will be given to the participant, and the informed consent process will be documented in the participant's research record. Consent with the participant's signature will serve as documentation. An opportunity will be provided to all potential participants for individual, private discussion of the study and the consent document before they sign the consent. All members of the research team will be trained and certified in participant consent procedures, the study protocol, human subjects protection, and HIPAA regulations.

Enrollment is expected to begin in Year 2 Quarter 3, and will remain open until recruitment goals are met, which is expected to be Year 4 Quarter 2.

4. Collect data. For each participant, participation will take place over 22 weeks (Weeks 1-4: Pre-intervention data collection; Weeks 5-16: Intervention; Weeks 17-22: Post-intervention data collection). Table 3 describes the study measures and outcomes. Data collection will take place at pre-intervention and post-intervention for each participant. At enrollment (i.e., preintervention) and one week after the 12th food box delivery (i.e. post-intervention), participants will provide data on glycemic control (measured by HbA1c), physical activity, body mass index (BMI), T2D self-management behaviors, T2D knowledge, T2D self-efficacy, and food security. To enhance the study's significance in characterizing the diet patterns and fruit and vegetable consumption of low-income food insecure people with T2D, we are collecting extensive diet quality data measures pre-intervention and post-intervention. Specifically, we will collect 24hour dietary recalls. Participants will be asked to document their dietary intake over a 24-hour period three times within four weeks. Two of the dietary recalls must be collected from a weekday and one of the recalls must be collected from a weekend day. Also, Skin carotenoid level will be measured using a Veggie Meter® optical skin scanner, which uses Raman Spectroscopy. The Veggie Meter assesses frequency changes in reflected light to calculate carotenoid presence. Skin carotenoid levels are a biomarker of fruit and vegetable dietary

PI: Krista Langston

*intake.* Participants will be asked to complete a survey via (email, text or in person) asking about their preference for the food provided in the food boxes.

Initial data collection will take place in a private space immediately following enrollment. The remaining pre-intervention data collection and post-intervention data collections will take place via telephone and at locations of each participant's choosing (e.g., HbA1c will be collected at home or at a community-based location such as a food pantry). Our team has necessary expertise and equipment to complete data collection in homes or community-based locations, having successfully completed thousands of such data collection events.<sup>37,43,54-61</sup>

The study has a single-arm, pre-post study design. All participants will receive the intervention (i.e., 12 weekly food boxes including the adapted DSME materials). Our target sample size for recruitment is 100. Assuming a repeated measures t-test, two-sided α=.05, and a Pearson correlation between repeated measures of r=.5, we will have 80% power to detect a Cohen's d effect size of 0.28. For context, Chrvala, Sherr, & Lipman's (2016) meta-analysis found that on average DSME led to a 0.6% improvement in HbA1c.<sup>25</sup> Assuming a standard deviation of 1.5%, this translates to Cohen's d of 0.4 (i.e., 0.6/1.5=0.4). Thus, the proposed intervention with a sample size of 100 is powered to detect a small-to-medium effect consistent with the expected effect size for standard DSME interventions in the context of research trials, and smaller than the effect found in previous food pantry-based DSME interventions.<sup>33,34</sup>

| Table 3. Delivering Health study measures and outcomes | |
|---|---|
| Variables | Instrument(s) or Measure(s) |
| <b>COVARIATES</b> | |
| Demographic | Demographic (age, gender, marital status, race, number of adults and |
| & | children in the household) and socioeconomic (education, employment |
| Socioeconomic | status, insurance coverage, WIC and SNAP benefits) variables will be |
| | captured using validated questions from the Behavior Risk Factor |
| | Surveillance System (BRFSS) <sup>62</sup> and National Health Interview Study |
| | (NHIS). <sup>120</sup> |
| EFFECTIVENESS OUTCOMES | |
| HbA1c | Finger stick blood collection will be used to test HbA1c using a Siemens |
| | DCA Vantage analyzer that can be taken into the field. <sup>63</sup> |
| Diet Quality | Skin carotenoid level will be measured using a Veggie Meter® optical skin |
| and Fruit and | scanner, which uses Raman Spectroscopy. The Veggie Meter assesses |
| Vegetable | frequency changes in reflected light to calculate carotenoid presence. |
| Consumption | |
| | 24-hour dietary recalls will be collected using the widely-used Nutrition |
| | Data System for Research (NDSR) software, which includes over 18,000 |
| | foods. <sup>64</sup> NDSR will be used to calculate Healthy Eating Index-2015 (HEI) |
| | scores and fruit and vegetable consumption. HEI-2015 scores comprise nine |

# PI: Krista Langston

| | component scores (e.g., vegetables, dairy) and are recommended by National Cancer Institute to assess impact of diet quality interventions. 65,66 |
|---|---|
| BMI | Weight and height will be used to compute a continuous measure of BMI |
| | using the Quetelet Index (kg/m <sup>2</sup> ). Weight will be measured in light clothing |
| | to the nearest 0.5 lb. (0.2 kg) using a calibrated digital scale. Height (without |
| | shoes) will be measured to the nearest 0.5 in. using a stadiometer. |
| Medical | BRFFS self-report items will assess lifetime prevalence of medical |
| Conditions | conditions. <sup>62</sup> |
| T2D Self- | The Summary of Diabetes Self-Care Activities (SDSCA) will be used to |
| Management | measure self-care activities. The SDSCA consists of 12 items to assess the |
| Behaviors | frequency of performing diabetes self-care tasks. <sup>67</sup> SDSCA was validated in |
| | minority populations, including the Marshallese. <sup>68</sup> |
| Oral Health | Oral health will be assessed by a single-item taken from the BRFFS |
| | survey. <sup>62</sup> |
| T2D Self- | Self-efficacy for health behaviors will be assessed through the Diabetes |
| Efficacy | Management Self-Efficacy Scale (DMSES), which assesses the extent to |
| | which respondents are confident in managing their blood sugar, diet, and |
| | exercise. <sup>69</sup> DMSES was validated in several studies of minority populations, |
| | including the Marshallese. <sup>68</sup> |
| T2D-related | Psychological distress related to type-2 diabetes will be assessed through |
| Distress | PAID-5 scale of the Diabetes Attitudes, Wishes, and Needs second study questionnaire (DAWN2) <sup>122</sup> |
| Food Security | Food security will be assessed using the adapted 10-item USDA screener. 121 |
| Food Pantry | Food pantry utilization will be assessed through modified items from Feeding America's |
| Utilization | Hunger in America Client Survey <sup>123</sup> |
| Medication | Measures of diabetes medication adherence will be collected with measures from BRFFS <sup>62</sup> , |
| Adherence | NHIS <sup>120</sup> , and ARMS-D. <sup>124</sup> |
| Coalrina Chilla | Aggregation of postion onto confidence in following a simple region and |
| Cooking Skills and | Assessment of participants confidence in following a simple recipe and cooking from basic ingredients will be assessed using items developed for |
| Knowledge | use in low socioeconomic populations. 125 |
| | LUATION MEASURES |
| Process | Process evaluation will include tracking indicators of retention (e.g., |
| Indicators | numbers of participants enrolled, data collection events completed) and |
| Indicators | numbers of participants enrolled, data collection events completed) and dosage (e.g., food boxes successfully received). Post-intervention data |
| Indicators | numbers of participants enrolled, data collection events completed) and dosage (e.g., food boxes successfully received). Post-intervention data collection will include open-ended questions about satisfaction with food |

## <u>5. Implement intervention.</u> **Table 4** summarizes the intervention.

Insecurity

PI: Krista Langston

| Table 4. DSM | Table 4. DSME and T2D-appropriate Food Boxes Intervention |
|---|---|
| | ■ Consistent with the American Association of Diabetes Educators, the adapted |
| <b>Evidence-</b> | ACP DSME will cover the topics of understanding diabetes, eating right, being |
| based | active, checking blood sugar, taking medicines, keeping feet healthy, and |
| DSME | insulin. The adapted curriculum consists of 12 modules, which will include |
| Curriculum | recipes and information on cooking and shopping when on a limited income and |
| | with foods commonly found at food pantries. |
| | ■ Each weekly food box will include ~9,000 calories of food, equivalent to the |
| T2D- | amount the average household receives <i>prorated per week</i> from an average |
| appropriate | Arkansas food pantry. <sup>37</sup> The boxes will follow the American Diabetes |
| food boxes | Association Create Your Plate method, consistent with the ACP DSME. Food |
| | will be purchased from a local grocery store. |
| | ■ Food boxes will be delivered to participants' homes once per week. Each |
| | week's box will include a two-page educational fact sheet version of the week's |
| Intervention | DSME module, including links and QR codes leading to videos supporting the |
| Delivery | week's curriculum module. Links to the week's online materials, which present |
| | the same content as the paper materials, will be texted or emailed to each |
| | participant the day their box is delivered. |
| Dosage | ■ 12 food boxes (including curriculum) delivered once per week over 12 weeks |

Given the study's longitudinal design, participant retention will be crucial. We engaged stakeholders to develop a retention plan. The plan specifies that study staff responsible for recruitment and retention will be bilingual (Spanish/English or Marshallese/English). Study staff will obtain each participant's contact information and preferred method of contact. Before each follow-up data collection visit or call, research staff will contact participants about the upcoming data collection.

"Participants will be offered a \$40 gift card for participation in each of the two data collection events for a total of \$80. Those participants who only participate in the survey or biometric data collection will receive \$20 for their time. Participants will also be offered \$10 gift cards at each of the dietary recall phone interviews for a total of \$60. Participants will only receive gift cards for the data collection events they complete. If a participant drops out, the study team will document who dropped out and why the drop out occurred. Participants will be able to choose a Tango electronic gift card at each of the data collection events.

## **Study Population**

Up to 110 study participants will be recruited from food pantries located in Benton and Washington Counties in northwest Arkansas.

## Inclusion Criteria

• 18 years of age or older

• Food insecure (confirmed with adapted 10-item screener)

• HbA1c levels of >7

Insecurity

PI: Krista Langston

## **Exclusion Criteria**

• Conditions making it unlikely the participant will be able to follow the protocol, such as terminal illness, non-ambulatory, severe mental illness, severely impaired vision or hearing, eating disorder, or plans to move out of the geographic region

- Pregnant
- Only one adult per household will be enrolled

#### **Risks and Benefits**

A risk to study participants is the potential for loss of confidentiality of study data. Measures to protect the confidentiality of study data will be implemented as described in the Data Handling and Recordkeeping section below.

A finger stick is required to collect a small amount of blood for testing, this may cause some discomfort.

The food box deliveries will be packaged to hold the correct temperature of perishable foods for three hours. After that time, or if the box is in any way damaged there is a risk of potentially eating spoiled foods from the food box delivery. There is also a risk of consuming a food item that the participant is unknowingly allergic to. We will do our best to ensure the integrity of the food box deliveries and are always available to contact with any questions regarding the food items in the deliveries.

Potential benefits include provision of nutritionally balanced food to participant's home for the 12 week period of the study. Participants may experience improved health status, specifically related to type 2 diabetes.

In addition to the potential of benefits to the participants, knowledge gained from the study could potentially benefit patients in the future.

## **Data Handling and Recordkeeping**

The Principal Investigator will carefully monitor study procedures to protect the safety of research subjects, the quality of the data and the integrity of the study.

All study subject material will be assigned a unique identifying code or number. The key to the code will be stored in a secure location in the Office of Community Health and Research. Only the principal investigator and the study coordinator will have access to the code and information that identifies the subject in this study. During data collection events survey data will be collected on a UAMS iPad or laptop using REDCap mobile app (with built in encryption technology). As soon as the data collectors return to UAMS, they will upload the data to the REDCap instance housed on a secure UAMS server and delete the data from the iPad or laptop. Blood specimens collected for HbA1c testing are only used for point of care testing, they will be discarded immediately after the test is performed. At the conclusion of the study the key to the code will be shredded, the data will be permanently de-identified.

PI: Krista Langston

The study will comply with UAMS Admin Guide Policy 3.2.01 – research data, reports and analyses be retained for seven years after final reporting or publication of a project, or longer if required by a sponsor or regulation.

## **Data Analysis**

Analyses will be performed with SAS 9.4. Data will be examined for distributional normality and outliers prior to analyses. Descriptive statistics will be generated for all variables of interest. We will examine patterns and predictors of missing values. If the percentage of missing values is larger than approximately 10%, we will compare models using multiple imputation with those using complete case analysis to examine the potential impact of missing values on the results.

To examine the intervention's effect on the primary outcomes of glycemic control as measured by HbA1c and diet quality as measured by Healthy Eating Index-2015 (HEI) scores, we will use mixed effects regression models for repeated measures. These analyses will focus on testing for a statistically significant difference between pre-intervention versus post-intervention measures. Additional analyses will include relevant covariates such as sex or age. We will also explore models that include process indicators of dosage of intervention received (e.g., number of food boxes received) to examine whether dosage predicts change in primary outcomes.

#### **Ethical Considerations**

This study will be conducted in accordance with all applicable government regulations and University of Arkansas for Medical Sciences research policies and procedures. This protocol and any amendments will be submitted and approved by the UAMS Institutional Review Board (IRB) to conduct the study.

The formal consent of each subject, using the IRB-approved consent form, will be obtained before that subject is submitted to any study procedure. All subjects for this study will be provided a consent form describing this study and providing sufficient information in language suitable for subjects to make an informed decision about their participation in this study. The person obtaining consent will thoroughly explain each element of the document and outline the risks and benefits, alternate treatment(s), and requirements of the study. The consent process will take place in a quiet and private room, and subjects may take as much time as needed to make a decision about their participation. Participation privacy will be maintained and questions regarding participation will be answered. No coercion or undue influence will be used in the consent process. This consent form must be signed by the subject and the person obtaining the consent. A copy of the consent will be given to the participant, and the informed consent process will be documented in the research record.

A \$40 Walmart gift card will be provided to the participant each time they complete a data collection event. If they complete both data collection events, they will receive a total of \$80 in Walmart gift cards.

#### **Dissemination of Data**

PI: Krista Langston

Results of this study may be used for presentations, posters, or publications. The publications will not contain any identifiable information that could be linked to a participant. The study will be listed on clinicaltrials.gov in accordance with funder requirements. A summary of results will be returned to participants in an infographic that is provided to them in person and/or mailed to the participants. After publication of the major findings in peer-reviewed journals, we will make the dataset available to other researchers for further analyses.

Version #: 10

Date: 20230222

IRB#260304

Page 11

PI: Krista Langston

## References

- 1. Centers for Disease Control and Prevention. *National Diabetes Statistics Report, 2017: Estimates of Diabetes and its Burden in the United States.* Atlanta, GA: Centers for Disease Control and Prevention, U.S. Dept of Health and Human Services;2017.
- 2. Rowley WR, Bezold C, Arikan Y, Byrne E, Krohe S. Diabetes 2030: Insights from Yesterday, Today, and Future Trends. *Popul Health Manag.* 2017;20(1):6-12.
- 3. Coleman-Jensen A, Rabbitt M, Gregory C, Singh A. *Household Food Security in the United States in 2017*. Washington, DC: U.S. Department of Agriculture, Economic Research Service:2018.
- 4. Gregory CA, Coleman-Jensen A. *Food Insecurity, Chronic Disease, and Health Among Working-Age Adults.* Washington, DC: United States Department of Agriculture, Economic Research Service;2017.
- 5. Centers for Disease Control and Prevention. BRFSS Prevalence & Trends Data. Centers for Disease Control and Prevention, National Center for Chronic Disease Prevention and Health Promotion, Division of Population Healh.

  https://www.cdc.gov/brfss/brfssprevalence/. Published 2019. Accessed February 1, 2019.
- 6. Gundersen C, Dewey A, Kato M, Crumbaugh A, Strayer M. Map the Meal Gap 2019: A Report on County and Congressional District Food Insecurity and County Food Cost in the United States in 2017. Chicago, IL: Feeding America;2019.
- 7. Seligman HK, Jacobs EA, Lopez A, Tschann J, Fernandez A. Food insecurity and glycemic control among low-income patients with type 2 diabetes. *Diabetes Care*. 2012;35(2):233-238.
- 8. Nguyen BT, Shuval K, Bertmann F, Yaroch AL. The Supplemental Nutrition Assistance Program, Food Insecurity, Dietary Quality, and Obesity Among U.S. Adults. *Am J Public Health*. 2015;105(7):1453-1459.
- 9. Berkowitz SA, Gao X, Tucker KL. Food-insecure dietary patterns are associated with poor longitudinal glycemic control in diabetes: results from the Boston Puerto Rican Health study. *Diabetes Care*. 2014;37(9):2587-2592.
- 10. Leung CW, Epel ES, Ritchie LD, Crawford PB, Laraia BA. Food insecurity is inversely associated with diet quality of lower-income adults. *J Acad Nutr Diet*. 2014;114(12):1943-1953.e1942.
- 11. Leung CW, Tester JM. The Association between Food Insecurity and Diet Quality Varies by Race/Ethnicity: An Analysis of National Health and Nutrition Examination Survey 2011-2014 Results. *J Acad Nutr Diet*. 2018;[Epub ahead of print]:e1-11.
- 12. Hanson KL, Connor LM. Food insecurity and dietary quality in US adults and children: a systematic review. *Am J Clin Nutr.* 2014;100(2):684-692.
- 13. Fram MS, Ritchie LD, Rosen N, Frongillo EA. Child experience of food insecurity is associated with child diet and physical activity. *J Nutr.* 2015;145(3):499-504.
- 14. To QG, Frongillo EA, Gallegos D, Moore JB. Household food insecurity is associated with less physical activity among children and adults in the U.S. population. *J Nutr*. 2014;144(11):1797-1802.
- 15. Leung C, Tester J, Laraia B. Household food insecurity and ideal cardiovascular health factors in U.S. adults. *JAMA Intern Med.* 2017;177(5):730-732.

## PI: Krista Langston

- 16. Berkowitz SA, Basu S, Meigs JB, Seligman HK. Food Insecurity and Health Care Expenditures in the United States, 2011-2013. *Health Serv Res.* 2018;53(3):1600-1620.
- 17. Choi SK, Fram MS, Frongillo EA. Very Low Food Security in US Households Is Predicted by Complex Patterns of Health, Economics, and Service Participation. *J Nutr.* 2017;147(10):1992-2000.
- 18. Kollannoor-Samuel G, Vega-Lopez S, Chhabra J, Segura-Perez S, Damio G, Perez-Escamilla R. Food insecurity and low self-efficacy are associated with health care access barriers among Puerto-Ricans with type 2 diabetes. *J Immigr Minor Health*. 2012;14(4):552-562.
- 19. American Diabetes Association. Standards of Medical Care in Diabetes 2019. *Diabetes Care*. 2019;42(Suppl 1):S1-S193.
- 20. Weinfield N, Mills G, Borger C, et al. *Hunger in America 2014: National Report Prepared for Feeding America*. Chicago, IL: Feeding America;2014.
- 21. Wetherill MS, Williams MB, White KC, Seligman HK. Characteristics of Households of People With Diabetes Accessing US Food Pantries: Implications for Diabetes Selfmanagement Education and Support. *Diabetes Educ.* 2019;[Epub ahead of print]:145721719857547.
- 22. Simmet A, Depa J, Tinnemann P, Stroebele-Benschop N. The Nutritional Quality of Food Provided from Food Pantries: A Systematic Review of Existing Literature. *J Acad Nutr Diet.* 2017;117(4):577-588.
- 23. Simmet A, Depa J, Tinnemann P, Stroebele-Benschop N. The Dietary Quality of Food Pantry Users: A Systematic Review of Existing Literature. *J Acad Nutr Diet*. 2017;117(4):563-576.
- 24. Powers MA, Bardsley J, Cypress M, et al. Diabetes Self-management Education and Support in Type 2 Diabetes: A Joint Position Statement of the American Diabetes Association, the American Association of Diabetes Educators, and the Academy of Nutrition and Dietetics. *Diabetes Care*. 2015;38(7):1372-1382.
- 25. Chrvala CA, Sherr D, Lipman RD. Diabetes self-management education for adults with type 2 diabetes mellitus: A systematic review of the effect on glycemic control. *Patient Educ Couns*. 2016;99(6):926-943.
- 26. Deakin T, McShane C, Cade JE, Williams RD. Group based training for self management startegies in people with type 2 diabetes mellitus. *Cochrane Database Syst Rev.* 2005;18(2):CD003417.
- 27. Steinsbekk A, Rygg LO, Lisulo M, Rise MB, Fretheim A. Group based diabetes self-management education compared to routine treatment for people with type 2 diabetes mellitus. A systematic review with meta-analysis. *BMC Health Serv Res.* 2012;12:213.
- 28. Tang TS, Funnell MM, Noorulla S, Oh M, Brown MB. Sustaining short-term improvements over the long-term: results from a 2-year diabetes self-management support (DSMS) intervention. *Diabetes Res Clin Pract.* 2012;95(1):85-92.
- 29. Baig A, Benitez A, Quinn M, Burnet D. Family interventions to improve diabetes outcomes for adults. *Ann N Y Acad Sci.* 2015;1353:89-112.
- 30. Robbins JM, Thatcher GE, Webb DA, Valdmanis VG. Nutritionist visits, diabetes classes, and hospitalization rates and charges: the Urban Diabetes Study. *Diabetes Care*. 2008;31(4):655-660.

## PI: Krista Langston

- 31. Healy SJ, Black D, Harris C, Lorenz A, Dungan KM. Inpatient diabetes education is associated with less frequent hospital readmission among patients with poor glycemic control. *Diabetes Care*. 2013;36(10):2960-2967.
- 32. Johnson TM, Murray MR, Huang Y. Associations between self-management education and comprehensive diabetes clinical care. *Diabetes Spectrum*. 2010;23(1):41-46.
- 33. Seligman HK, Lyles C, Marshall MB, et al. A pilot food bank intervention featuring diabetes-appropriate food improved glycemic control among clients in three states. *Health Aff (Millwood)*. 2015;34(11):1956-1963.
- 34. Seligman HK, Smith M, Rosenmoss S, Marshall MB, Waxman E. Comprehensive diabetes self-management support from food banks: a randomized controlled trial. *Am J Public Health*. 2018;108(9):1227-1234.
- 35. Yeary KHK, Long CR, Bursac Z, McElfish PA. Design of a randomized controlled comparative effectiveness trial testing a Family Model of Diabetes Self-Management Education (DSME) vs. standard DSME for Marshallese in the United States. *Contemp Clin Trials Commun.* 2017;6:97-104.
- 36. Yeary KH, Aitaoto N, Sparks K, et al. Cultural Adaptation of Diabetes Self-Management Education for Marshallese Residing in the United States: Lessons Learned in Curriculum Development. *Prog Community Health Partnersh.* 2017;11(3):253-261.
- 37. Long CR, Rowland B, McElfish PA. Intervention to improve access to fresh fruits and vegetables among Arkansas food pantry clients. *Prev Chronic Dis.* 2019;16:E09.
- 38. Long CR, Rowland B, Langston K, et al. Reducing the Intake of Sodium in Community Settings: Evaluation of Year One Activities in the Sodium Reduction in Communities Program, Arkansas, 2016-2017. *Prev Chronic Dis.* 2018;15:E160.
- 39. Kennedy BM, Champagne CM, Ryan DH, et al. The "Rolling Store:" an economical and environmental approach to the prevention of weight gain in African American women. *Ethn Dis.* 2009;19(1):7-12.
- 40. Palar K, Napoles T, Hufstedler LL, et al. Comprehensive and medically appropriate food support is associated with improved HIV and diabetes health. *J Urban Health*. 2017;94(1):87-99.
- 41. Flynn MM, Reinert S, Schiff AR. A six-week cooking program of plant-based recipes improves food security, body weight, and food purchases for food pantry clients. *J Hunger Environ Nutr.* 2013;8(1):73-84.
- 42. Hixson L, Hepler B, Kim M. *The Native Hawaiian and Other Pacific Islander population 2010*. Washington, DC: United States Census Bureau;2012.
- 43. McElfish P, Rowland B, Long C, et al. Diabetes and hypertension in Marshallese adults: Results from faith-based health screenings. *J Racial Ethn Health Disparities*. 2017;4(6):1042-1050.
- 44. Galinsky A, Zelaya C, Simile C, Barnes P. *Health conditions and behaviors of Native Hawaiian and Pacific Islander persons in the United States, 2014.* Hyattsville, MD: National Center for Health Statistics;2017.
- 45. Karter AJ, Schillinger D, Adams AS, et al. Elevated rates of diabetes in Pacific Islanders and Asian subgroups The Diabetes Study of Northern California (DISTANCE). *Diabetes Care*. 2013;36(3):574-579.

## PI: Krista Langston

- 46. Mau MK, Sinclair K, Saito EP, Baumhofer KN, Kaholokula JK. Cardiometabolic health disparities in Native Hawaiians and other Pacific Islanders. *Epidemiol Rev.* 2009;31:113-129.
- 47. Wallace AS, Seligman HK, Davis TC, et al. Literacy-appropriate educational materials and brief counseling improve diabetes self-management. *Patient Educ Couns*. 2009;75(3):328-333.
- 48. American College of Physicians. *Living with Diabetes: An Everyday Guide for You and Your Family.* Philadelphia, PA: American College of Physicians;2017.
- 49. American Diabetes Association. Create Your Plate. American Diabetes Association. <a href="http://www.diabetes.org/food-and-fitness/food/planning-meals/create-your-plate/">http://www.diabetes.org/food-and-fitness/food/planning-meals/create-your-plate/</a>. Published 2019. Accessed July 9, 2019.
- 50. Feeding America. Foods to Encourage Background. Feeding America. <a href="http://hungerandhealth.feedingamerica.org/wp-content/uploads/legacy/mp/files/tool\_and\_resources/files/f2e-background-detail.v1.pdf">http://hungerandhealth.feedingamerica.org/wp-content/uploads/legacy/mp/files/tool\_and\_resources/files/f2e-background-detail.v1.pdf</a>. Published 2015. Accessed February 5, 2019.
- 51. US Department of Agriculture, US Department of Health and Human Services. *Dietary Guidelines for Americans*, 2010. Washington, DC: US Department of Agriculture;2010.
- 52. US Department of Health and Human Services, US Department of Agriculture. 2015-2020 Dietary Guidelines for Americans, 8th ed. Washington, DC: US Department of Health and Human Services;2015.
- 53. United States Department of Agriculture. *U.S. Adult Food Security Survey Module: Three-Stage Design, with Screeners*. Washington, DC: USDA, Economic Research Service;2012.
- 54. McElfish P, Bridges M, Hudson J, et al. Family model of diabetes education with a Pacific Islander community. *Diabetes Educ.* 2015;41(6):706-715.
- 55. Donoho G, McElfish P, Avants R, Hallgren E. A novel recruiting and surveying method: participatory research during a Pacific Islander community's traditional cultural event. *Gateways: International Journal of Community Research and Engagement.* 2015:8(1):150-159.
- 56. McElfish PA, Goulden PA, Bursac Z, et al. Engagement practices that join scientific methods with community wisdom: designing a patient-centered, randomized control trial with a Pacific Islander community. *Nurs Ing.* 2017;24(2):1-11.
- 57. McElfish PA, Long CR, Kaholokula JK, et al. Design of a comparative effectiveness randomized controlled trial testing a faith-based Diabetes Prevention Program (WORD DPP) vs. a Pacific culturally-adapted Diabetes Prevention Program (PILI DPP) for Marshallese in the United States. *Medicine*. 2018;97(19):e0677.
- 58. McElfish PA, Long CR, Selig JP, et al. Health Research Participation, Opportunity, and Willingness Among Minority and Rural Communities of Arkansas. *Clin Transl Sci.* 2018;11(5):487-497.
- 59. McElfish P, Long C, Kohler P, et al. Comparative effectiveness and maintenance of diabetes self-management education interventions for Marshallese type 2 diabetes patients: a randomized controlled trial. *Diabetes Care*. 2019;42:1-9.
- 60. Felix H, Rowland B, Long CR, et al. Diabetes Self-Care Behaviors Among Marshallese Adults Living in the United States. *J Immigr Minor Health*. 2018;20(6):1500-1507.

## PI: Krista Langston

- 61. Ayers BL, Shreve MD, Scott AL, et al. Social and economic influences on infant and child feeding practices in a Marshallese community. *Public Health Nutr*. 2019;22(8):1461-1470.
- 62. Centers for Disease Control and Prevention. Behavioral Risk Factor Surveillance System (BRFSS). http://www.cdc.gov/brfss/. Published 2017. Accessed May 28, 2018, 2018.
- 63. Lenters-Westra E, Slingerland RJ. Six of eight hemoglobin A1c point-of-care instruments do not meet the general accepted analytical performance criteria. *Clin Chem*. 2010;56(1):44-52.
- 64. University of Minnesota. NDSR Software. University of Minnesota Nutrition Coordinating Center. <a href="http://www.ncc.umn.edu/products/">http://www.ncc.umn.edu/products/</a>. Published 2019. Accessed July 7, 2019.
- 65. Krebs-Smith SM, Pannucci TE, Subar AF, et al. Update of the Healthy Eating Index: HEI-2015. *J Acad Nutr Diet*. 2018;118(9):1591-1602.
- 66. Reedy J, Lerman JL, Krebs-Smith SM, et al. Evaluation of the Healthy Eating Index-2015. *J Acad Nutr Diet*. 2018;118(9):1622-1633.
- 67. Toobert DJ, Hampson SE, Glasgow RE. The summary of diabetes self-care activities measure: results from 7 studies and a revised scale. *Diabetes Care*. 2000;23(7):943-950.
- 68. Bohanny W, Wu S, Liu C, Yeh S, Tsay S, Wang T. Health literacy, self-efficacy, and self-care behaviors in patients with type 2 diabetes mellitus. *Journal Of The American Association Of Nurse Practitioners*. 2013;25(9):495-502.
- 69. Bijl JV, Poelgeest-Eeltink AV, Shortridge-Baggett L. The psychometric properties of the diabetes management self-efficacy scale for patients with type 2 diabetes mellitus. *J Adv Nurs.* 1999;30(2):352-359.
- 70. Long CR, Stewart MK, Cunningham TV, Warmack TS, McElfish PA. Health research participants' preferences for receiving research results. *Clinical Trials*. 2016;13(6):582-591
- 71. Long CR, Stewart MK, McElfish PA. Health research participants are not receiving research results: a collaborative solution is needed. *Trials*. 2017;18(1):449.
- 72. Long C, Purvis R, Flood-Grady E, et al. Health researchers' experiences, perceptions, and barriers related to sharing study results with participants. *Health Research Policy and Systems*. 2019;17(25).
- 73. Rowland B, Mayes K, Faitak B, Stephens RM, Long CR, McElfish PA. Improving Health while Alleviating Hunger: Best Practices of a Successful Hunger Relief Organization. *Curr Dev Nutr.* 2018;2(9):nzy057.
- 74. Hunger Solutions Minnesota, SuperShelf. *2017 Minnesota Food Shelf Client Survey*. Minneapolis, MN: University of Minnesota, SuperShelf;2018.
- 75. An R, Wang J, Liu J, Shen J, Loehmer E, McCaffrey J. A systematic review of food pantry-based interventions in the USA. *Public Health Nutr.* 2019;22(9):1704-1716.
- 76. Simmet A, Stroebele-Benschop N. Creating healthy food pantries by using behavioural economics approaches. *Public Health Nutr.* 2019:1-3.
- 77. Remley D, Gallagher T, McDowell J, Kershaw M, Lambea M, Melgar-Quinonez H. Extension's role in developing "choice" food pantries in southwest Ohio. *J Extension*. 2006;44(6):6IAW5.
- 78. Remley DT, Kaiser ML, Osso T. A case study of promoting nutrition and long-term food security through choice pantry development. *J Hunger Environ Nutr.* 2013;8(3):324-336.

## PI: Krista Langston

- 79. Stluka S, Moore L, Eicher-Miller HA, et al. Voices for food: methodologies for implementing a multi-state community-based intervention in rural, high poverty communities. *BMC Public Health*. 2018;18(1):1055.
- 80. Byker Shanks C. Promoting Food Pantry Environments that Encourage Nutritious Eating Behaviors. *J Acad Nutr Diet*. 2017;117(4):523-525.
- 81. Caspi CE, Canterbury M, Carlson S, et al. A behavioural economics approach to improving healthy food selection among food pantry clients. *Public Health Nutr.* 2019; [Epub ahead of print]:1-11.
- 82. United States Department of Agriculture. SNAP-Ed Library. USDA, SNAP-Ed Connection. https://snaped.fns.usda.gov/library. Published 2019. Accessed July 8, 2019.
- 83. Feeding America. Resources. Feeding America.

  <a href="https://hungerandhealth.feedingamerica.org/resources/">https://hungerandhealth.feedingamerica.org/resources/</a>. Published 2019. Accessed July 7, 2019.
- 84. Feldman M, Schwartz MB. *A Tipping Point: Leveraging Opportunities to Improve the Nutritional Quality of Food Bank Inventory.* Los Angeles, CA: MAZON;2018.
- 85. Mousa TY, Freeland-Graves JH. Impact of food pantry donations on diet of a low-income population. *Int J Food Sci Nutr.* 2019;70(1):78-87.
- 86. Martin KS, Wu R, Wolff M, Colantonio AG, Grady J. A novel food pantry program: food security, self-sufficiency, and diet-quality outcomes. *Am J Prev Med.* 2013;45(5):569-575.
- 87. Chapnick M, Barnidge E, Sawicki M, Elliott M. Healthy options in food pantries a qualitative analysis of factors affecting the provision of healthy food items in St. Louis, Missouri. *J Hunger Environ Nutr.* 2019;14(1-2):262-280.
- 88. Wetherill MS, Williams MB, White KC, Li J, Vidrine JI, Vidrine DJ. Food pantries as partners in population health: assessing organizational and personnel readiness for delivering nutrition-focused charitable food assistance. *J Hunger Environ Nutr.* 2019;14(1-2):50-69.
- 89. Bryan AD, Ginsburg ZA, Rubinstein EB, et al. Foods and Drinks Available from Urban Food Pantries: Nutritional Quality by Item Type, Sourcing, and Distribution Method. *J Community Health.* 2019;44(2):339-364.
- 90. Wilson NL, Just DR, Swigert J, Wansink B. Food pantry selection solutions: a randomized controlled trial in client-choice food pantries to nudge clients to targeted foods. *J Public Health (Oxf)*. 2017;39(2):366-372.
- 91. Remley DT, Zubieta AC, Lambea MC, Quinonez HM, Taylor C. Spanish- and English-speaking client perceptions of choice food pantries. *J Hunger Environ Nutr.* 2010;5(1):120-128.
- 92. Remley D, Franzen-Castle L, McCormack L, Eicher-Miller HA. Chronic health condition influences on client perceptions of limited or non-choice food pantries in low-income, rural communities. *Am J Health Behav.* 2019;43(1):105-118.
- 93. Martin KS, Colantonio AG, Picho K, Boyle KE. Self-efficacy is associated with increased food security in novel food pantry program. *SSM Popul Health*. 2016;2:62-67.
- 94. Booth S, Begley A, Mackintosh B, et al. Gratitude, resignation and the desire for dignity: lived experience of food charity recipients and their recommendations for improvement, Perth, Western Australia. *Public Health Nutr.* 2018;21(15):2831-2841.

## PI: Krista Langston

- 95. The Ohio Association of Second Harvest Foodbanks. Making the Switch: A Guide for Converting to a Client Choice Food Pantry. The Ohio Association of Second Harvest Foodbanks. <a href="http://ohiofoodbanks.org/docs/publications/ChoicePantryGuide.pdf">http://ohiofoodbanks.org/docs/publications/ChoicePantryGuide.pdf</a>. Published 2009. Accessed April 26, 2019.
- 96. Cooksey-Stowers K, Read M, Wolff M, Martin KS, McCabe M, Schwartz M. Food pantry staff attitudes about using a nutrition rating system to guide client choice. *J Hunger Environ Nutr.* 2019;14(1-2):35-49.
- 97. Hadden KB, Arnold CL, Curtis LM, et al. Rationale and development of a randomized pragmatic trial to improve diabetes outcomes in patient-centered medical homes serving rural patients. *Contemp Clin Trials*. 2018;73:152-157.
- 98. Glasgow RE, Vogt TM, Boles SM. Evaluating the public health impact of health promotion interventions: the RE-AIM framework. *Am J Public Health*. 1999;89(9):1322-1327.
- 99. McElfish P, Long C, Rowland B, Moore S, Wilmoth R, Ayers B. Improving culturally appropriate care using a community-based participatory approach: evaluation of a multi-component cultural competency training program, Arkansas, 2015-2016. *Prev Chronic Dis.* 2017;14(E26).
- 100. McElfish PA, Moore R, Buron B, et al. Integrating Interprofessional Education and Cultural Competency Training to Address Health Disparities. *Teach Learn Med*. 2018;30(2):213-222.
- 101. McNeill C, Washburn L, Hadden KB, Moon Z. Evaluating the Effectiveness of the How to Talk to Your Doctor HANDbook Program. *Health Lit Res Pract*. 2019;3(2):e103-e109.
- 102. Haller J, Keller Z, Barr S, Hadden K, Oliphant SS. Assessing Readability: Are Urogynecologic Patient Education Materials at an Appropriate Reading Level? *Female Pelvic Med Reconstr Surg.* 2019;25(2):139-144.
- 103. Prince LY, Schmidtke C, Beck JK, Hadden KB. An Assessment of Organizational Health Literacy Practices at an Academic Health Center. *Qual Manag Health Care*. 2018;27(2):93-97.
- 104. McElfish P, Rowland B, Ayers B, et al. Development and evaluation of a community-engaged research training program: building capacity of Marshallese stakeholders and academic researchers to conduct health research. *Gateways*. 2019;12(1):1-20.
- 105. Mykerezi E, Mills B. The impact of food stamp program participation on household food insecurity. *Am J Agric Econ.* 2010;92(5):1379-1391.
- 106. Berkowitz SA, Seligman HK, Choudhry NK. Treat or eat: food insecurity, cost-related medication underuse, and unmet needs. *Am J Med.* 2014;127(4):303-310.e303.
- 107. Kinsey E, Dupuis R, Oberle M, Hillier A, Cannuscio C. Chronic Disease Self-Management During the Monthly SNAP Cycle (P04-193-19). *Curr Dev Nutr.* 2019;3(Suppl 1).
- 108. Ippolito MM, Lyles CR, Prendergast K, Marshall MB, Waxman E, Seligman HK. Food insecurity and diabetes self-management among food pantry clients. *Public Health Nutr.* 2017;20(1):183-189.
- 109. Food Research & Action Center. *Addressing Food Insecurity: A Toolkit for Pediatricians*. Washington, DC: Food Research & Action Center, American Academy of Pediatrics;2017.

## PI: Krista Langston

- 110. Smith S, Malinak D, Chang J, Schultz A, Brownell K. Addressing Food Insecurity in Family Medicine and Medical Education. *Fam Med.* 2017;49(10):765-771.
- 111. Bickley LS. *Bates' Pocket Guide to Physical Examination and History Taking*. 8th ed. Philadelphia, PA: Wolters Kluwer; 2017.
- 112. Cox CL. *Physical Assessment for Nurses and Healthcare Professionals*. 3rd ed. Hoboken, NJ: John Wiley & Sons; 2019.
- 113. Aspry KE, Van Horn L, Carson JAS, et al. Medical Nutrition Education, Training, and Competencies to Advance Guideline-Based Diet Counseling by Physicians: A Science Advisory From the American Heart Association. *Circulation*. 2018;137(23):e821-e841.
- 114. Patil SP, Craven K, Kolasa K. Food Insecurity: How You Can Help Your Patients. *Am Fam Physician*. 2018;98(3):143-145.
- 115. Frank JR, Snell LS, Cate OT, et al. Competency-based medical education: theory to practice. *Med Teach*. 2010;32(8):638-645.
- 116. Carraccio C, Englander R, Van Melle E, et al. Advancing Competency-Based Medical Education: A Charter for Clinician-Educators. *Acad Med.* 2016;91(5):645-649.
- 117. Sierpina VS, Welch K, Devries S, et al. What Competencies Should Medical Students Attain in Nutritional Medicine? *J Nutr Food Sci.* 2015;5(6):1000431.
- 118. American Hospital Association. *Social Determinants of Health Series: Food Insecurity and the Role of Hospitals.* Chicago, IL: Health Research & Educational Trust;2017.
- 119. National Academy of Medicine. *Strategic Plan 2018-2023: Goalposts for a Healthier Future*. Washington, DC: National Academy of Medicine;2017.
- 120. Centers for Disease Control and Prevention. National Health Interview Study (NHIS). https://www.cdc.gov/nchs/nhis/2020nhis.htm. Published 2020. Accessed March 22, 2021.
- 121. Hager, E. R., Quigg, A. M., Black, M. M., Coleman, S. M., Heeren, T., Rose-Jacobs, R., ... & Frank, D. A. (2010). Development and validity of a 2-item screen to identify families at risk for food insecurity. Pediatrics, 126(1), e26-e32.
- 122. Nicolucci A, Kovacs Burns K, Holt RI, Comaschi M, Hermanns N, Ishii H, Kokoszka A, Pouwer F, Skovlund SE, Stuckey H, Tarkun I, Vallis M, Wens J, Peyrot M; DAWN2 Study Group. Diabetes Attitudes, Wishes and Needs second study (DAWN2<sup>TM</sup>): crossnational benchmarking of diabetes-related psychosocial outcomes for people with diabetes. Diabet Med. 2013;30(7):767-77. doi: 10.1111/dme.12245
- 123. America, F. (2014). Hunger in America 2014. National Report. August.
- 124. Kripalani, S., Risser, J., Gatti, M. E., & Jacobson, T. A. (2009). Development and evaluation of the Adherence to Refills and Medications Scale (ARMS) among low-literacy patients with chronic disease. Value in Health, 12(1), 118-123.
- 125. Frans, N. (2017). Development of cooking skills questionnaire for EFNEP participants in Kansas (Doctoral dissertation, Kansas State University).